CLINICAL TRIAL: NCT02280317
Title: A Phase I/II, Dose Escalation Study To Assess The Safety and Tolerability of VAL201 In Patients With Advanced or Metastatic Prostate Cancer and Other Advanced Solid Tumours
Brief Title: Dose Finding Safety Study of VAL201 in Cancer Patients
Acronym: VAL201-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ValiRx Plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VAL201-001; 2013-004009-25 (EudraCT Number)
Record Dates: First submitted 2014-10-20; First posted 2014-10-31 (Estimated); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Stage III Prostate Carcinoma; Stage IV Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose Escalation sequential assignment
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1: 0.5 mg/kg (Experimental): VAL201-001 Sub-cutaneous injection. 0.5 mg/kg
  Interventions: Drug: VAL201
- Cohort 2: 1 mg/kg (Experimental): VAL201-001 Sub-cutaneous injection. 1.0 mg/kg
  Interventions: Drug: VAL201
- Cohort 3: 2 mg/kg (Experimental): VAL201-001 Sub-cutaneous injection. 2.0 mg/kg
  Interventions: Drug: VAL201
- Cohort 4: 4 mg/kg (Experimental): VAL201-001 Sub-cutaneous injection. 4.0 mg/kg
  Interventions: Drug: VAL201
- Cohort 5: up to 8 mg/kg (Experimental): VAL201-001 Sub-cutaneous injection. 8.0 mg/kg; potential to escalate to 16 mg/kg after 3 cycles according to clinician decision Flexibility of dosing enabled under protocol.
  Interventions: Drug: VAL201

INTERVENTIONS:
Drug: VAL201 — VAL201-001 Sub-cutaneous injection.
  Other Names: VAL201-001

SUMMARY:
Dose finding safety study of VAL201 in cancer patients.

DETAILED DESCRIPTION:
A Phase I/II, dose escalation study to assess the safety and tolerability of VAL201 in patients with locally advanced or metastatic prostate cancer and other advanced solid tumours.

ELIGIBILITY:
The study will enrol patients with locally advanced or metastatic prostate cancer. The MTD/MAD may also be evaluated in patients with other advanced tumour types for whom no standard effective therapy is available and a rationale for use of VAL201 exists.

The average timeframe is 18-26 weeks per subject and the outcome measured is a composite average for each group.

* Inclusion criteria:

  * Specific Inclusion Criteria for Patients with Prostate Cancer
  * Patients with incurable, locally advanced or metastatic prostate cancer where a policy of intermittent hormone therapy has been decided. Who have specific clinical parameters.
* Specific Inclusion Criteria for Patients with Other Advanced Solid Tumours

  * Patients with histologically and/or cytologically confirmed advanced solid tumour for whom no standard effective therapy is available and a rationale for use of VAL201 exists.
  * Patients with incurable, locally advanced or metastatic prostate cancer where a policy of intermittent hormone therapy has been decided. These patients must also have the following:

    1. Rising PSA on three samples (once non-castrate levels established); each over 2 weeks apart, with the last two values being greater than 2 ng/mL. Higher than and at least 25% over the nadir.
    2. Absent or very mild prostate cancer-related symptoms.
    3. No plans for any therapy for prostate cancer in the next two months.
  * General Inclusion Criteria for all Patients
  * Adult patients defined by age greater than 18 years at time of consent.
  * Ability to give written, informed consent prior to any study-specific Screening procedures, with the understanding that the consent may be withdrawn by the patient at any time without prejudice.
  * Patient is capable of understanding the protocol requirements, is willing and able to comply with the study protocol procedures, and has signed the informed consent document.
  * Evaluable disease, either measurable on imaging, or with informative tumour marker(s) and a set of specific biochemical and haematological parameters relating to the specific cancer.
  * Negative human chorionic gonadotropin (hCG) test in women of childbearing potential.
  * Sexually active male and female patients of childbearing potential must agree to use an effective method of birth control. Female patients may be surgically sterile.
  * Laboratory values at Screening:

    * Absolute neutrophil count ≥1.5 x 109/L.
    * Platelets ≥100 x 109/L.
    * Haemoglobin ≥9 g/dL without blood transfusion or colony stimulating factor support.
    * Total bilirubin <1.5 times the upper limit of normal (ULN);
    * AST (SGOT) ≤2.5 times the ULN;
    * ALT (SGPT) ≤2.5 times the ULN; ≤5 x ULN for patients with advanced solid tumours with liver metastases.
    * Serum creatinine ≤1.5 x ULN or estimated glomerular filtration rate (GFR) of >50 mL/min based on the Cockcroft-Gault formula.
* Exclusion criteria

  * Specific Exclusion Criteria for Patients with Prostate Cancer Patients has received an anticancer therapy, including investigational agents, within the precious 6 weeks or 4 weeks.
  * Any patients who have undergone prior orchidectomy.
  * Specific Exclusion Criteria for Patients with Other Advanced Solid Tumours Pregnant or lactating female patients.
  * Documented, symptomatic or uncontrolled brain metastases.
  * History of clinically significant cardiac condition, including ischemic cardiac event, myocardial infarction or unstable cardiac disease within 3 months previous to the indication of home therapy.
  * Known Human Immunodeficiency Virus positivity.
  * Active Hepatitis B or C or other active liver disease (other than malignancy).
  * Any active, clinically significant, viral, bacterial, or systemic fungal infection within previous 4 weeks prior to home therapy.
  * Any medical history that would jeopardize compliance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study will enrol patients with locally advanced or metastatic prostate cancer. The MTD/MAD may also be evaluated in patients with other advanced tumour types for whom no standard effective therapy is available and a rationale for use of VAL201 exists.
Pre-assignment Details: Interventional Study Model; Sequential Assignment
  -Dose Escalation sequential assignment-
Groups:
- Cohort 1: 0.5 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection 0.5mg/kg.
- Cohort 2: 1.0 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection 1.0 mg/kg.
- Cohort 3: 2.0 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection 2.0 mg/kg
- Cohort 4: 4.0 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection 4.0 mg/kg
- Cohort 5: Up to 8.0 mg/kg: VAL201-001 Sub-cutaneous injection. 8.0 mg/kg; potential to escalate to 16 mg/kg after 3 cycles according to clinician decision Flexibility of dosing enabled under protocol.
Period: Overall Study
Arm/Group | Cohort 1: 0.5 mg/kg | Cohort 2: 1.0 mg/kg | Cohort 3: 2.0 mg/kg | Cohort 4: 4.0 mg/kg | Cohort 5: Up to 8.0 mg/kg
Started | 1 (Patients receiving at least one dose.) | 1 (Patients receiving at least one dose.) | 3 (Patients receiving at least one dose.) | 5 (Patients receiving at least one dose.) | 2 (Patients receiving at least one dose.)
Completed | 1 (Patients completing six cycles.) | 1 (Patients completing six cycles.) | 0 (Patients completing six cycles.) | 2 (Patients completing six cycles.) | 0 (Patients completing six cycles.)
Not Completed | 0 | 0 | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: 0.5 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection 0.5 mg/kg.
- Cohort 2: 1 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection 1.0 mg/kg.
- Cohort 3: 2 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection 2.0 mg/kg.
- Cohort 4: 4 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection 4.0 mg/kg.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 0.5 mg/kg | Cohort 2: 1 mg/kg | Cohort 3: 2 mg/kg | Cohort 4: 4 mg/kg | Cohort 5: up to 8 mg/kg | Total
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 2 | 12
Age, Continuous [Mean (Full Range); unit: years] | 70 [70 to 70] | 62 [62 to 62] | 76 [69 to 81] | 72.6 [60 to 84] | 73 [71 to 75] | 72.4 [60 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 3 | 5 | 2 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 1 | 1 | 2 | 4 | 2 | 10
  Race/Ethnicity: Black/African American | 0 | 0 | 1 | 0 | 0 | 1
  Race/Ethnicity: Asian | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1 | 1 | 3 | 5 | 2 | 12
Stage of Cancer at Screening [Count of Participants; unit: Participants]
  Metastatic Prostate Cancer | 1 | 0 | 1 | 2 | 1 | 5
  Locally Advanced Prostate Cancer | 0 | 1 | 2 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose-Limiting Toxicity
Description: The number of Dose-Limiting Toxicity events is used to determine whether a maximum tolerated dose (MTD) is obtained.
Time Frame: The average timeframe is 18-26 weeks per subject
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 0.5 mg/kg | Cohort 2: 1.0 mg/kg | Cohort 3: 2.0 mg/kg | Cohort 4: 4.0 mg/kg | Cohort 5: up to 8 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 2
Participants
  Dose-limiting Toxicity observed (DLT) | 0 | 0 | 0 | 0 | 1
  Dose-reduction required | 0 | 0 | 0 | 0 | 0
  MTD or MAD proposed | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics of VAL201. (Cmax)
Description: Assessment of pharmacokinetic variables at multiple time points (5 min, 10 min, 15 min, 30 min, 60 min, 90 min, 2 hours, 3 hours, 4 hours, 6 hours and 8 hours after dosing) and multiple dosing days (Cycle 1 Day 1, Cycle 3 Day 1, Cycle 4 Day 1 and Cycle 6 Day 1) for each patient analysed.
Time Frame: The average timeframe is 18-26 weeks per subject
Population: Cohort 5 consisted of one participant dosed at 8 mg/kg and one participant dosed at 4 mg/kg, on which pharmacokinetic parameters were measured; pharmacokinetic data was not analysed for Cohorts 1-4. Pharmacokinetic profiles were collected on multiple dosing days.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Cohort 5: up to 8.0 mg/kg: VAL201 Sub-cutaneous injection. 8.0 mg/kg
- Cohort 5: up to 8 mg/kg: VAL201 Sub-cutaneous injection 4 mg/kg
Arm/Group | Cohort 5: up to 8.0 mg/kg | Cohort 5: up to 8 mg/kg
Number analyzed (Participants) | 1 | 1
ng/mL | 3323 [2522 to 4232] | 2205 [1448 to 2765]

3. Secondary Outcome: Pharmacokinetics of VAL201 (AUC 0-inf)
Description: as for outcome 2
Time Frame: The average timeframe is 18-26 weeks per subject
Population: as for outcome 2
Measure: Mean (Full Range); unit: ug/mL*h
Groups:
- Cohort 5: up to 8 mg/kg AUC: VAL201 Sub-cutaneous injection 8.0 mg/kg
- Cohort 5: Up to 8 mg/kg: VAL201 Sub-cutaneous injection 4.0 mg/kg
Arm/Group | Cohort 5: up to 8 mg/kg AUC | Cohort 5: Up to 8 mg/kg
Number analyzed (Participants) | 1 | 1
ug/mL*h | 5.0 [4.78 to 5.28] | 3.8 [2.36 to 4.51]

4. Other Pre Specified Outcome: Number of Patients Who Completed 6 Cycles of Treatment
Description: The number of patients who completed 6 cycles of treatment is compared with the number who withdrew prior to completion of the scheduled 6 cycles
Time Frame: The average timeframe is 18-26 weeks per subject
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 5: up to 8.0 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection. 8.0 mg/kg; potential to escalate to 16 mg/kg after 3 cycles according to clinician decision.
  Flexibility of dosing enabled under protocol.
Arm/Group | Cohort 1: 0.5 mg/kg | Cohort 2: 1.0 mg/kg | Cohort 3: 2.0 mg/kg | Cohort 4: 4.0 mg/kg | Cohort 5: up to 8.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 2
Participants
  Completed 6 cycles of treatment | 1 | 1 | 0 | 1 | 1
  Withdrew from trial prior to completion | 0 | 0 | 3 | 4 | 1

5. Other Pre Specified Outcome: Number of Patients Displaying Disease Progression by PCWG2 and/or RECIST Criteria
Description: Assessment of disease response to treatment by PCWG2 and/or RECIST. Disease progression is defined by RECIST 1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; and by PCWG2 criteria that PSA values did not see an increase of 25% or more and absolute increase of 2 ng/mL or more from the nadir.
Time Frame: The average timeframe is 18-26 weeks per subject
Population: Excludes one participant from Cohort 4 who received a single dose
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 5: up to 8.0 mg/kg: VAL201: VAL201-001 Sub-cutaneous injection. 8.0 mg/kg; potential to escalate to 16 mg/kg after 3 cycles according to clinician decision Flexibility of dosing enabled under protocol.
Arm/Group | Cohort 1: 0.5 mg/kg | Cohort 2: 1.0 mg/kg | Cohort 3: 2.0 mg/kg | Cohort 4: 4.0 mg/kg | Cohort 5: up to 8.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 4 | 2
Participants
  Showed no progressive disease during trial period according to PCWG2 | 1 | 0 | 1 | 3 | 1
  Showed progressive disease at any point during trial period according to PCWG2 | 0 | 1 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: 18 weeks.
Description: All events experienced by patients recorded here, regardless of assessment of causality as related or not to drug treatment. Cohort 5 has been segregated into Cohort 5 (8 mg/kg) and Cohort 5 (4 mg/kg) to delineate the actual dose given in this group.
Groups:
- Cohort 5: up to 8 mg/kg (8 mg/kg): VAL201-001 Sub-cutaneous injection. 8.0 mg/kg; potential to escalate to 16 mg/kg after 3 cycles according to clinician decision Flexibility of dosing enabled under protocol.
  This patient received 8 mg/kg
- Cohort 5: up to 8 mg/kg (4 mg/kg): VAL201-001 Sub-cutaneous injection. 8.0 mg/kg; potential to escalate to 16 mg/kg after 3 cycles according to clinician decision Flexibility of dosing enabled under protocol.
  This patient received 4 mg/kg
Arm/Group | Cohort 1: 0.5 mg/kg | Cohort 2: 1.0 mg/kg | Cohort 3: 2.0 mg/kg | Cohort 4: 4.0 mg/kg | Cohort 5: up to 8 mg/kg (8 mg/kg) | Cohort 5: up to 8 mg/kg (4 mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 0/5 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 2/5 | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 5/5 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 0.5 mg/kg (N=1) | Cohort 2: 1.0 mg/kg (N=1) | Cohort 3: 2.0 mg/kg (N=3) | Cohort 4: 4.0 mg/kg (N=5) | Cohort 5: up to 8 mg/kg (8 mg/kg) (N=1) | Cohort 5: up to 8 mg/kg (4 mg/kg) (N=1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 0.5 mg/kg (N=1) | Cohort 2: 1.0 mg/kg (N=1) | Cohort 3: 2.0 mg/kg (N=3) | Cohort 4: 4.0 mg/kg (N=5) | Cohort 5: up to 8 mg/kg (8 mg/kg) (N=1) | Cohort 5: up to 8 mg/kg (4 mg/kg) (N=1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hot Flushes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site brusing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Finger deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"There is an agreement in place with the PI and the sponsor that restricts the PI's rights to discuss and publish the trial results after the trial is completed".

DOCUMENTS (3):
  • Study Protocol (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT02280317/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT02280317/SAP_001.pdf
  • Informed Consent Form (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT02280317/ICF_002.pdf